CLINICAL TRIAL: NCT01077804
Title: Fifteen Year Follow-up to Evaluate Long-term Effectiveness of VARIVAX Among Children and Adolescents
Brief Title: A Study to Evaluate Long-term Impact of VARIVAX Among Children and Adolescents (V210-036)(COMPLETED)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Kaiser Permanente (Other)
Responsible Party: Sponsor
Other Study IDs: V210-036; 2010_014 (Other: Merck); EP08005.002 (Other: Merck)
Record Dates: First submitted 2010-02-26; First posted 2010-03-01 (Estimated); Results first posted 2011-11-03 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-08

CONDITIONS: Varicella; Herpes Zoster
MeSH Terms: conditions — Chickenpox; Herpes Zoster

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Varivax vaccinated children: Children who are members of Kaiser Permanente Medical Care Program (KPMCP) and who received a first dose of the varicella vaccine, Varivax, in 1995 between the ages of 12 and 23 months.

SUMMARY:
The purpose of these continuing post-licensure studies is to evaluate the long-term effectiveness of VARIVAX® [Varicella Virus Vaccine Live (Oka/Merck)] and to assess the impact of the vaccine on the epidemiology of varicella and herpes zoster.

DETAILED DESCRIPTION:
Parents/guardians of the cohort of children vaccinated between 12 and 23 months of age during a six-month period in 1995 (June-November) at KPMCP Northern California were interviewed by telephone at 6-month intervals to ascertain whether their child had varicella or herpes zoster in the 6 months prior to interview. Follow-up continued for a minimum of 14 years after vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Subject was a member of Kaiser Permanente Northern California, age 12-23 months, received a dose of varicella vaccine between June and November 1995, and parents accepted to participate in 15-year follow-up

Exclusion Criteria:

* Subjects diagnosed with varicella before study enrollment
* Subject's parents unable to complete telephone interviews in English, Spanish, or Cantonese

Ages: 12 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 15 years prospective follow-up of the original study cohort
Sampling Method: Probability Sample
Enrollment: 7585 (Actual)
Dates: Start 1995-06-01 (Actual); Primary Completion 2010-09-01 (Actual); Study Completion 2010-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger Baxter, Principal Investigator — Kaiser Permanente

REFERENCES:
- [Result] Baxter R, Ray P, Tran TN, Black S, Shinefield HR, Coplan PM, Lewis E, Fireman B, Saddier P. Long-term effectiveness of varicella vaccine: a 14-Year, prospective cohort study. Pediatrics. 2013 May;131(5):e1389-96. doi: 10.1542/peds.2012-3303. Epub 2013 Apr 1. PMID 23545380

RESULTS

PARTICIPANT FLOW:
Groups:
- Varivax Vaccinated Children: Children who are members of Kaiser Permanente Medical Care Program (KPMCP) and who received a first dose (0.5 mL) of the varicella vaccine, Varivax, in 1995 between the ages of 12 and 23 months.
Period: Overall Study
Arm/Group | Varivax Vaccinated Children
Started | 7585
Completed | 7386
Not Completed | 199
Not completed — Unreachable | 102
Not completed — Refused to continue | 79
Not completed — Other | 18

BASELINE CHARACTERISTICS:
Arm/Group | Varivax Vaccinated Children
Number analyzed (Participants) | 7585
Age, Customized [Number; unit: Participants] | 7585
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3714
  Male | 3871
Region of Enrollment [Number; unit: participants]
  United States | 7585

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants With an Occurrence of Herpes Zoster Infection
Description: Herpes zoster cases were physician-diagnosed cases.
Time Frame: From 6 weeks to 168 months (14 years) post vaccination
Measure: Number; unit: Participants
Arm/Group | Varivax Vaccinated Children
Number analyzed (Participants) | 7585
Participants | 46

2. Primary Outcome: Number of Participants With an Occurrence of Breakthrough Varicella
Description: Parents/guardians of Varivax vaccinated children were interviewed every 6 months after vaccination. The number of participants with varicella (referred to as varicella with "any symptoms") were reported by parents during the interview. No medical confirmation of the diagnosis was required.
Time Frame: From 6 weeks to 168 months (14 years) post vaccination
Measure: Number; unit: Participants
Arm/Group | Varivax Vaccinated Children
Number analyzed (Participants) | 7585
Participants
  Any Varicella symptoms | 1425
  Varicella with >50 lesions | 362
  Varicella with >300 lesions | 28

3. Primary Outcome: Incidence Rate of Breakthrough Varicella
Description: as for outcome 2
Time Frame: From 6 weeks to 168 months (14 years) post vaccination
Measure: Number (95% Confidence Interval); unit: Rate per 1000 person years
Arm/Group | Varivax Vaccinated Children
Number analyzed (Participants) | 7585
Rate per 1000 person years
  Any varicella | 15.9 [15.1 to 16.7]
  Varicella with > 50 lesions | 4 [3.6 to 4.9]
  Varicella with > 300 lesions | 0.3 [0.2 to 0.5]

4. Secondary Outcome: Incidence Rate of Herpes Zoster Infection
Description: Herpes zoster cases were physician-diagnosed.
Time Frame: From 6 weeks to 168 months (14 years) post vaccination
Measure: Number (95% Confidence Interval); unit: Rate per 1000 person years
Arm/Group | Varivax Vaccinated Children
Number analyzed (Participants) | 7585
Rate per 1000 person years | 0.45 [0.33 to 0.60]

ADVERSE EVENTS:
Description: The purpose of this study was to monitor changes in vaccine effectiveness over time and no collection of adverse events was required. Therefore, no data on adverse events were collected and the number at risk is zero.
Arm/Group | Varivax Vaccinated Children
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission, it being understood that the results of this study are not to be considered confidential. The sponsor review can be expedited to meet publication guidelines.